CLINICAL TRIAL: NCT01064076
Title: S-ICD® System Clinical Investigation
Brief Title: S-ICD® System IDE Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DN-03909
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2015-07

CONDITIONS: Tachycardia, Ventricular
Keywords: ICD, defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-ICD System (Experimental): This is a single arm study
  Interventions: Device: S-ICD System

INTERVENTIONS:
Device: S-ICD System — The S-ICD System is an implantable technology that uses a subcutaneous pulse generator and subcutaneous electrode system to treat ventricular tachyarrhythmias. The S-ICD System consists of the SQ-RX pulse generator (Model 1010), the Q-TRAK subcutaneous electrode (Model 3010), the Q-TECH programmer (Model 2020), and Q-GUIDE electrode insertion tools (Models 4010 and 4020).
  Other Names: SQ-RX Pulse Generator; Q-TRAK Subcutaneous Electrode; Q-GUIDE Electrode Insertion Tools; Q-TECH Programmer

SUMMARY:
This clinical study is designed to evaluate the safety and effectiveness of the subcutaneous implantable defibrillator (S-ICD) System.

DETAILED DESCRIPTION:
This clinical study is a prospective, non-randomized, multicenter clinical study without a control group conducted in the United States, Europe, and New Zealand.

Patients meeting eligibility criteria for implanting an S-ICD System will be enrolled in this clinical study, implanted with an S-ICD System, and followed prior to hospital discharge, and post-implant at 30 days, 90 days, and 180 days. After the 180-day post-implant follow-up visit, patients will continue to be followed semi-annually until study closure.

Eligible patients enrolled in this clinical study may also participate in the chronic conversion sub-study.

The safety endpoint will be evaluated through the use of a 180-day S-ICD System complication-free rate. The effectiveness endpoint will be evaluated using an induced ventricular fibrillation (VF) conversion efficacy rate. Spontaneous episodes and chronic conversion testing data will be evaluated using descriptive statistics to provide additional data supporting the continued chronic performance of the S-ICD System.

ELIGIBILITY:
Inclusion Criteria:

* For patients without an existing transvenous device

  • Patient meets Class I, Class IIa or Class IIb indications/recommendations for ICD implantation per the current published guidelines at the time of enrollment
* For patients with an existing transvenous device

  • Patient requires replacement or revision of an existing implanted transvenous ICD system
* Age is ≥ 18 years
* An appropriate pre-operative ECG per template provided

Exclusion Criteria:

* Any condition which precludes the subject's ability to comply with the study requirements, including completion of the study.
* Females who are pregnant or lactating and pre-menopausal women who are unwilling to use adequate birth control for the duration of the study.
* Participation in any other investigational study without prior written consent from the study sponsor.
* Patients with a serious medical condition and life expectancy of less than one year.
* Patients with documented spontaneous and frequently recurring VT that is reliably terminated with anti-tachycardia pacing, unless the patient is not a candidate for a transvenous ICD system.
* Patients with existing epicardial patches or subcutaneous electrodes in the left thoracic quadrant.
* Patients with unipolar pacemakers or implanted devices that revert to unipolar pacing.
* Patients with severely impaired kidney function as measured by a Cockcroft-Gault Glomerular Filtration Rate (GFR) with an estimated GFR ≤ 29.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Husby, M.S., MPH, Study Director — Cameron Health, Inc. a Subsidiary of Boston Scientific
Locations (33):
- United States (28):
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - Foothill Cardiology, Pasadena, California
  - CMCA / Sequoia Hospital, Redwood City, California
  - Sharp Grossmont Hospital, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Pacific Heart Institute, Santa Monica, California
  - South Bay Electrophysiology, Torrance, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Midwest Heart Foundation, Oakbrook Terrace, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Cooper University Hospital, Camden, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Mid Carolina Cardiology Research, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Heart Hospital, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Heart Clinics Northwest, Spokane, Washington
  - The Vancouver Clinic, Vancouver, Washington
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Papworth Hospital NHS Trust, Papworth Everard, Cambridge, United Kingdom

REFERENCES:
- [Derived] Amin AK, Gold MR, Burke MC, Knight BP, Rajjoub MR, Duffy E, Husby M, Stahl WK, Weiss R. Factors Associated With High-Voltage Impedance and Subcutaneous Implantable Defibrillator Ventricular Fibrillation Conversion Success. Circ Arrhythm Electrophysiol. 2019 Apr;12(4):e006665. doi: 10.1161/CIRCEP.118.006665. PMID 30917689
- [Derived] Burke MC, Gold MR, Knight BP, Barr CS, Theuns DAMJ, Boersma LVA, Knops RE, Weiss R, Leon AR, Herre JM, Husby M, Stein KM, Lambiase PD. Safety and Efficacy of the Totally Subcutaneous Implantable Defibrillator: 2-Year Results From a Pooled Analysis of the IDE Study and EFFORTLESS Registry. J Am Coll Cardiol. 2015 Apr 28;65(16):1605-1615. doi: 10.1016/j.jacc.2015.02.047. PMID 25908064
- [Derived] Weiss R, Knight BP, Gold MR, Leon AR, Herre JM, Hood M, Rashtian M, Kremers M, Crozier I, Lee KL, Smith W, Burke MC. Safety and efficacy of a totally subcutaneous implantable-cardioverter defibrillator. Circulation. 2013 Aug 27;128(9):944-53. doi: 10.1161/CIRCULATIONAHA.113.003042. PMID 23979626
- See also: Boston Scientific Website — http://www.bostonscientific.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 33 investigational sites participated in the study, twenty-eight (28) of which were in the United States, 2 in New Zealand, 2 in The Netherlands and 1 in the United Kingdom. A total of 330 patients were enrolled between January 27, 2010 and May 20, 2011.
Pre-assignment Details: Of the 330 enrollments, 321 underwent an implant procedure (implant attempt) and 9 were withdrawn prior to the commencement of the implant procedure.
Period: Overall Study
Arm/Group | S-ICD System
Started | 321 (321 subjects underwent an implant procedure for the S-ICD System)
Completed | 303 (303 subjects completed a minimum of 180 days of follow up)
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: All patients with an attempted implant of the S-ICD System.
Arm/Group | S-ICD System
Number analyzed (Participants) | 321
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 253
  >=65 years | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 238
Region of Enrollment [Number; unit: participants]
  United States | 275
  Netherlands | 16
  United Kingdom | 1
  New Zealand | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free of Type I Complications at 180 Days.
Description: Percentage of Participants Free of Type I Complications at 180 days compared to the performance goal of 79%. Type I complications are those caused by the S-ICD System.
Time Frame: 180 days
Population: The analysis cohort includes all subjects undergoing an implant attempt.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Single Arm: Cohort includes all subjects undergoing an implant attempt
Arm/Group | Single Arm
Number analyzed (Participants) | 321
percentage of participants | 99.0 [97.9 to NA] — This was a one-sided CI

2. Primary Outcome: Percentage of Participants Who Pass Induced VF Conversion Test
Description: Percentage of participants who pass induced VF conversion test was compared to a performance goal of 88%. Definition of a success was two consecutive successful 65 joule shocks out of four attempts in the same polarity.
Time Frame: Implant/Pre-Discharge
Population: 304 subjects had a complete VF conversion test recorded
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | S-ICD System
Number analyzed (Participants) | 304
percentage of participants | 96.5 [93.8 to 98.2]

ADVERSE EVENTS:
Arm/Group | S-ICD System
Serious Adverse Events (participants affected / at risk) | 52/321
Other Adverse Events (participants affected / at risk) | 104/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-ICD System (N=321)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute Appendicitis (Blood and lymphatic system disorders) | 1 (1)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adverse Reaction to Medication (Surgical and medical procedures) | 4 (4)
Angina (Cardiac disorders) | 1 (1)
Bleeding (Surgical and medical procedures) | 1 (1)
Erosioin (Skin and subcutaneous tissue disorders) | 3 (3)
GI Disorder (Gastrointestinal disorders) | 3 (3)
Heart Failure/Worsening of Heart Failure (Cardiac disorders) | 10 (15)
Hyponatremia (General disorders) | 1 (1)
Inability to Communicate with the Device (General disorders) | 1 (1)
Inappropriate Shock: Oversensing (General disorders) | 3 (3)
Inappropriate Shock: SVT Above Discrimination Zone (Normal Device Function) (General disorders) | 2 (2)
Incomplete Electrode Connection to the Device (General disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 5 (5)
Near Syncope/Dizziness/Shortness of Breath/Confusion (General disorders) | 2 (2)
Pancreatitis (General disorders) | 1 (1)
Pneumonia (General disorders) | 1 (1)
Pneumothorax (General disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Sub-optimal Electrode Position (General disorders) | 1 (1)
Suspected Device Malfunction (General disorders) | 1 (1)
Syncope (General disorders) | 2 (2)
Device System Infection - Explant (General disorders) | 4 (4)
VT Below Conditional Zone (General disorders) | 1 (1)
Worsening of Benign Prostatic Hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Worsening of VT/VF (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-ICD System (N=321)
Adverse Reaction to Medication (Surgical and medical procedures) | 4 (4)
Atrial Fibrillation/Flutter (Cardiac disorders) | 17 (17)
Discomfort (General disorders) | 23 (27)
Hematoma (Surgical and medical procedures) | 5 (6)
Inadequate/Prolonged Healing of Incision Site (Surgical and medical procedures) | 5 (5)
Inappropriate Shock (General disorders) | 45 (64)
Incision/Superficial Infection (Infections and infestations) | 15 (15)
Phantom Shock (General disorders) | 4 (6)
Suboptimal Pulse Generator and/or Electrode Position (Surgical and medical procedures) | 4 (4)
Syncope (General disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The major limitation of this study is the lack of a control group and the relatively short follow-up time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No